CLINICAL TRIAL: NCT00881751
Title: A Randomized Open-Label Multi-Institution Phase II Study of the Combination of Bevacizumab and Erlotinib Compared to Sorafenib in the First-Line Treatment of Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Bevacizumab and Erlotinib or Sorafenib as First-Line Therapy in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101282; MUSC-101282; GENENTECH-AVF4481s
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2015-10

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab; Erlotinib Hydrochloride; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: bevacizumab and erlotinib (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28.
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride
- Arm 2: sorafenib tosylate (Active Comparator): Patients receive oral sorafenib tosylate twice daily on days 1-28.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Arms: Arm 1: bevacizumab and erlotinib
Drug: erlotinib hydrochloride — Given orally
  Arms: Arm 1: bevacizumab and erlotinib
Drug: sorafenib tosylate — Given orally
  Arms: Arm 2: sorafenib tosylate

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib and sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Bevacizumab, erlotinib, and sorafenib may also stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether giving bevacizumab together with erlotinib is more effective than giving sorafenib in treating patients with liver cancer.

PURPOSE: This randomized phase II trial is studying how well giving bevacizumab together with erlotinib works compared with sorafenib as first-line therapy in treating patients with advanced liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the overall survival in patients with advanced hepatocellular carcinoma treated with bevacizumab and erlotinib hydrochloride vs sorafenib tosylate.

Secondary

* To estimate the event-free survival and tumor response rate of these patients.
* To evaluate the safety and tolerability of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28.
* Arm II: Patients receive oral sorafenib tosylate twice daily on days 1-28. In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed advanced hepatocellular carcinoma (HCC)

  * Childs-Pugh class A
  * CLIP score ≤ 5
* Not a candidate for curative surgical resection or loco-regional therapy
* Measurable disease as per RECIST 1.1 criteria, defined as ≥ 1 previously unirradiated, bidimensionally measurable lesion ≥ 20 mm by CT scan or MRI (triphasic spiral CT scan or MRI employing a "liver protocol" image capture technique required)

  * Bone lesions, ascites, and pleural effusions are not considered measurable lesions
* No fibrolamellar HCC
* No known brain metastases
* No prior organ transplantation

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 9 g/dL
* Transaminases ≤ 5 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 times ULN
* PT ≤ 1.8 times ULN

  * Prolonged INR allowed for patients who require full dose anticoagulation
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 45 mL/min
* Urine protein < 2+ by urine dipstick OR urine protein ≤ 1 g by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 weeks after completion of study treatment
* Able to take and absorb oral medication
* No active infection requiring parenteral therapy
* No known HIV or AIDS
* No uncontrolled blood pressure (BP), defined as systolic BP ≥ 150 mm Hg and/or diastolic BP ≥ 100 mm Hg
* No uncontrolled or significant cardiovascular disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Uncontrolled angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Grade 3 cardiac valve dysfunction
  * Cardiac arrhythmia not controlled by medication
  * Stroke or transient ischemic attack within the past 6 months
  * Arterial thrombotic event of any type within the past 6 months
* No significant or symptomatic vascular disease (e.g., aortic aneurysm, aortic dissection, or peripheral vascular disease) within the past 6 months
* No decompensated liver disease as evidenced by clinically significant ascites refractory to diuretic therapy, hepatic encephalopathy, or coagulopathy not corrected by conservative measures
* No grade 3 bleeding esophageal or gastric varices within the past 2 months

  * Prior variceal bleeding allowed provided patient has undergone banding or sclerotherapy and there has been no evidence of bleeding for 2 months
* No gastric varices ≥ grade 2
* No hemoptysis (i.e., ≥ ½ teaspoon of bright red blood per episode) within the past month
* No evidence of bleeding diathesis or coagulopathy
* No concurrent uncontrolled illness, including, but not limited to, a history of or current evidence of unexplained nephrotic syndrome or other severe illness/disease that would preclude study participation
* No history of hypertensive crisis or hypertensive encephalopathy
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious, non-healing wound, active ulcer, or untreated bone fracture
* No significant traumatic injury within the past 28 days
* No history of allergy to bevacizumab, erlotinib hydrochloride, sorafenib tosylate, or related compounds
* No other primary malignancy within the past 5 years, except carcinoma in situ of the cervix or urinary bladder or nonmelanoma skin cancer
* No mental incapacitation or psychiatric illness that would preclude study participation
* Not incarcerated or compulsorily detained (i.e., involuntarily incarcerated) for treatment of either a psychiatric or physical illness (e.g., infectious disease)

PRIOR CONCURRENT THERAPY:

* Prior surgery, local ablation, trans-arterial hepatic artery embolization, or trans-arterial chemoembolization are allowed provided the lesion(s) have progressed since treatment OR there are additional measurable, untreated lesions present
* No prior systemic therapy for HCC
* No prior organ transplantation
* More than 7 days since prior minor surgical procedures, fine needle aspirations, or core biopsies (excluding placement of a vascular access device)
* More than 28 days since any prior therapy
* More than 28 days since prior and no concurrent major surgical procedure or open biopsy
* More than 28 days since prior and no concurrent participation in another experimental drug study
* No other concurrent anticancer or antitumor therapy, including chemotherapy, radiotherapy, immunotherapy, or hormonal anticancer therapy
* No other concurrent investigational agents
* No concurrent warfarin (other types of anticoagulation allowed)

Ages: 18 Years to 116 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-03; Primary Completion 2016-05 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Columbia University/ New York Presbyterian Hospital, New York, New York
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, PLLCat Sarah Cannon Cancer Center, Nashville, Tennessee
  - UVA Cancer Center, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Subjects who were enrolled to the Bevacizumab + Erlotinib Arm.
  Bevacizumab: IV on days 1 and 15 of a 28 day cycle Erlotinib: Oral on days 1-28 of a 28 day cycle
- Arm II: Subjects who were enrolled to the sorafenib arm.
  Sorafenib: oral administration on days 1-28 of a 28 day cycle
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 47 | 48
Completed | 47 | 43
Not Completed | 0 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Any subjects who were enrolled to either Arm 1 or Arm 2
Groups:
- Arm I: Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28.
  bevacizumab: Given IV
  erlotinib hydrochloride: Given orally
- Arm II: Patients receive oral sorafenib tosylate twice daily on days 1-28.
  sorafenib tosylate: Given orally
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 27 | 56
  >=65 years | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 38 | 33 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 38 | 41 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 4 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 28 | 32 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment day 1 until death from any cause. Patients still alive at the end of follow up,patients who withdrew consent from the trial and patients who were lost to follow up will have their survival time censored at the last date of contact.
Time Frame: from date of day 1 until the date of death
Population: Only subjects who received one dose of study drug were considered for this outcome. 5 subjects enrolled to Arm II did not receive any study drug and were not evaluable for this outcome.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm I: Subjects who were enrolled to the Bevacizumab + Erlotinib Arm and received at least one dose of study drug.
  Bevacizumab: IV on days 1 and 15 of a 28 day cycle Erlotinib: Oral on days 1-28 of a 28 day cycle
- Arm II: Subjects who were enrolled to the sorafenib arm and received at least one dose of study drug.
  Sorafenib: oral administration on days 1-28 of a 28 day cycle
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 47 | 43
Months | 8.55 [7.00 to 13.9] | 8.55 [5.69 to 12.2]

2. Secondary Outcome: Event-free Survival
Description: EFS is defined as the time from randomization to any of the following three types of events: 1 - progression; 2 - withdrawal due to excessive toxicity; 3 - any other clinical event requiring withdrawal from the study.
Time Frame: From the time of randomization until progression, withdrawal due to toxicity or any other clinical event requiring withdrawal from the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 47 | 43
Months | 4.37 [2.99 to 7.36] | 2.76 [1.84 to 4.80]

3. Secondary Outcome: Number of SAEs Experienced
Description: The study will report the number of SAEs experienced in each arm. All patients who receive any study drug will be evaluable for toxicity.
Time Frame: From day 1 of drug administration until 30 days after the last dose of study drug.
Population: Patients who received at least one dose of study drug were included in this analysis.
Measure: Number; unit: serious adverse events
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 47 | 43
serious adverse events | 48 | 39

4. Secondary Outcome: Response Rate
Description: Secondary outcome measures include response rate as assessed on restaging imaging studies utilizing RECIST 1.1.
Time Frame: From day 1 drug administration until 30 days after the last dose of study drug.
Population: Responders include complete and partial responders defined by RECIST 1.1 criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 47 | 43
percentage of participants | 15 | 9

ADVERSE EVENTS:
Time Frame: From initiation of study drug administration until 30 days after last study drug administration
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 25/47 | 19/43
Other Adverse Events (participants affected / at risk) | 47/47 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=47) | Arm II (N=43)
cardiac arest (Cardiac disorders) | 2 (2) | 0 (0)
atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
esophageal varices hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
GI hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
esophageal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
septic arthritis (Infections and infestations) | 1 (1) | 0 (0)
osteomyelitis (Infections and infestations) | 2 (2) | 0 (0)
subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
encephalopathy (Nervous system disorders) | 3 (4) | 3 (3)
altered mental status (Nervous system disorders) | 1 (1) | 3 (3)
confusion (Nervous system disorders) | 0 (0) | 2 (2)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
rash (zoster) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
esophageal varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
fever (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1)
hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
lower extremity edema (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=47) | Arm II (N=43)
tinnitus (Ear and labyrinth disorders) | 2 | 3
anemia (Blood and lymphatic system disorders) | 0 | 3
hemoglobin (Blood and lymphatic system disorders) | 20 | 13
neutrophils (NOS) (Investigations) | 6 | 3
platelets (Blood and lymphatic system disorders) | 18 | 17
RBC decrease (Blood and lymphatic system disorders) | 0 | 2
WBC decrease (Blood and lymphatic system disorders) | 7 | 7
WBC increase (Blood and lymphatic system disorders) | 1 | 3
hypotension (Cardiac disorders) | 4 | 4
tachycardia (Cardiac disorders) | 0 | 2
hypertension (Cardiac disorders) | 20 | 14
INR (Investigations) | 3 | 2
chills (General disorders) | 14 | 7
dizziness (General disorders) | 5 | 12
fatigue (General disorders) | 33 | 33
fever (General disorders) | 15 | 5
headache (General disorders) | 7 | 6
hemorrhage (NOS) (General disorders) | 4 | 1
insomnia (General disorders) | 10 | 7
sweating (General disorders) | 1 | 4
weight loss (General disorders) | 25 | 17
weight gain (General disorders) | 0 | 2
acne (Skin and subcutaneous tissue disorders) | 27 | 4
alopecia (Skin and subcutaneous tissue disorders) | 13 | 9
blisters (Skin and subcutaneous tissue disorders) | 0 | 2
bruising (Skin and subcutaneous tissue disorders) | 0 | 3
dry skin (Skin and subcutaneous tissue disorders) | 24 | 17
erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 6
hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5 | 7
nail changes (Skin and subcutaneous tissue disorders) | 10 | 0
nail loss (Skin and subcutaneous tissue disorders) | 1 | 3
petechiae (Skin and subcutaneous tissue disorders) | 4 | 3
pruritus (Skin and subcutaneous tissue disorders) | 25 | 2
rash (Skin and subcutaneous tissue disorders) | 16 | 11
skin pain (Skin and subcutaneous tissue disorders) | 2 | 2
skin peeling (Skin and subcutaneous tissue disorders) | 0 | 2
skin redness (Skin and subcutaneous tissue disorders) | 0 | 2
abdominal pain (Gastrointestinal disorders) | 24 | 10
anorexia (Gastrointestinal disorders) | 29 | 19
ascites (Gastrointestinal disorders) | 9 | 1
bloating (Gastrointestinal disorders) | 1 | 2
constipation (Gastrointestinal disorders) | 6 | 11
dehydration (Gastrointestinal disorders) | 12 | 5
diarrhea (Gastrointestinal disorders) | 31 | 33
discolored stool (Gastrointestinal disorders) | 3 | 1
distension (Gastrointestinal disorders) | 3 | 3
dry mouth (Gastrointestinal disorders) | 15 | 4
dysgeusia (Gastrointestinal disorders) | 21 | 9
dyspepsia (Gastrointestinal disorders) | 11 | 3
dysphagia (Gastrointestinal disorders) | 6 | 3
flatulence (Gastrointestinal disorders) | 8 | 5
hemorrhoids (Gastrointestinal disorders) | 3 | 1
mucositis/stomatitis (NOS) (Gastrointestinal disorders) | 13 | 2
nausea (Gastrointestinal disorders) | 24 | 18
stomach pain (Gastrointestinal disorders) | 2 | 3
vomiting (Gastrointestinal disorders) | 12 | 17
encephalopathy (Hepatobiliary disorders) | 4 | 3
jaundice (Hepatobiliary disorders) | 1 | 2
edema (NOS) (General disorders) | 3 | 0
edema: limb (General disorders) | 7 | 14
edema: trunk (General disorders) | 0 | 2
albumin (NOS) (Metabolism and nutrition disorders) | 4 | 2
alkaline phosphatase (Metabolism and nutrition disorders) | 18 | 10
ALT (Metabolism and nutrition disorders) | 17 | 11
AST (Metabolism and nutrition disorders) | 25 | 13
bicarbonate decrease (Metabolism and nutrition disorders) | 1 | 2
bilirubin (Metabolism and nutrition disorders) | 21 | 13
BUN increase (Metabolism and nutrition disorders) | 1 | 3
calcium (NOS) (Metabolism and nutrition disorders) | 0 | 2
creatinine increase (Metabolism and nutrition disorders) | 6 | 5
Creatinine (NOS) (Metabolism and nutrition disorders) | 4 | 2
glucose (NOS) (Metabolism and nutrition disorders) | 3 | 2
hyperammonemia (Metabolism and nutrition disorders) | 1 | 2
hyperglycemia (Metabolism and nutrition disorders) | 8 | 7
hyperkalemia (Metabolism and nutrition disorders) | 6 | 0
hypermagnesemia (Metabolism and nutrition disorders) | 1 | 2
hypernatremia (Metabolism and nutrition disorders) | 3 | 1
hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 7
hypocalcemia (Metabolism and nutrition disorders) | 9 | 8
hypoglycemia (Metabolism and nutrition disorders) | 2 | 2
hypokalemia (Metabolism and nutrition disorders) | 11 | 5
hypomagnesemia (Metabolism and nutrition disorders) | 8 | 6
hyponatremia (Metabolism and nutrition disorders) | 15 | 12
hypophosphatemia (Metabolism and nutrition disorders) | 9 | 8
magnesium (NOS) (Metabolism and nutrition disorders) | 0 | 2
phosphorus (NOS) (Metabolism and nutrition disorders) | 0 | 2
potassium (NOS) (Metabolism and nutrition disorders) | 0 | 2
back pain (Musculoskeletal and connective tissue disorders) | 11 | 10
body ache (Musculoskeletal and connective tissue disorders) | 1 | 2
chest pain (Musculoskeletal and connective tissue disorders) | 4 | 7
extremity cramping (Musculoskeletal and connective tissue disorders) | 1 | 2
extremity pain (Musculoskeletal and connective tissue disorders) | 2 | 4
joint pain (Musculoskeletal and connective tissue disorders) | 8 | 7
muscle cramping (Musculoskeletal and connective tissue disorders) | 3 | 3
muscle pain (Musculoskeletal and connective tissue disorders) | 9 | 4
muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
shoulder pain (Musculoskeletal and connective tissue disorders) | 3 | 2
weakness (Musculoskeletal and connective tissue disorders) | 5 | 14
altered mental status (Psychiatric disorders) | 2 | 3
anxiety (Psychiatric disorders) | 5 | 3
ataxia (Nervous system disorders) | 1 | 2
confusion (Psychiatric disorders) | 5 | 4
depression (Psychiatric disorders) | 7 | 6
memory impairment (Nervous system disorders) | 1 | 2
sensory neuropathy (Nervous system disorders) | 3 | 4
syncope (Nervous system disorders) | 0 | 2
voice changes (Nervous system disorders) | 11 | 6
blurred vision (Eye disorders) | 1 | 2
dry eye (Eye disorders) | 9 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 14 | 6
dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 7
dysuria (Renal and urinary disorders) | 1 | 2
hematuria (Renal and urinary disorders) | 3 | 0
proteinuria (Renal and urinary disorders) | 14 | 7
urinary frequency/urgency (Renal and urinary disorders) | 8 | 1
urinary tract infection (Renal and urinary disorders) | 4 | 4
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 3
flu-like syndrome (General disorders) | 7 | 2
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes